CLINICAL TRIAL: NCT01702259
Title: A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of the Erchonia Scanner Device (GLS) Green Diode on Reducing the Appearance of Cellulite Clinical Study Protocol.
Brief Title: Study of the Effect of Low Level Laser Light Therapy on Reducing the Appearance of Cellulite in the Thighs and Buttocks.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMCTE002
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia Scanner device (GLS) (Experimental): The Erchonia® GLS device is made up of six independent diodes, each emitting 17 milliwatts (mW), 532 nanometer (nm) of green laser light.
  Interventions: Device: Erchonia Scanner device (GLS)
- Placebo device (Sham Comparator): Inactive Erchonia GLS device
  Interventions: Device: Placebo device

INTERVENTIONS:
Device: Erchonia Scanner device (GLS) — The Erchonia® GLS device is made up of six independent diodes, each emitting 17 milliwatts (mW), 532 nanometer (nm) of green laser light.
  Arms: Erchonia Scanner device (GLS)
Device: Placebo device — Inactive Erchonia GLS.
  Arms: Placebo device

SUMMARY:
The purpose of this study is to determine whether the application of green diode low level laser light therapy is effective in reducing the appearance of cellulite in the thighs and buttocks.

DETAILED DESCRIPTION:
Cellulite is a common term used to describe superficial pockets of trapped fat, which causes uneven dimpling or "orange peel" skin. It appears in 90% of post-adolescent women. In advanced stages of cellulite, heaviness and pain may occur.

Currently available treatments for cellulite have minimal to no demonstrable effect and some involve risky invasive procedures. Therefore, the potential advantages of the application of low level laser light therapy to reduce the appearance of cellulite over current treatment options include a risk free procedure that is non-invasive and pain free. Since low level laser light within the green spectrum has been proven to increase the synthesis of collagen, it is believed that its application may serve to decrease the appearance of cellulite by tightening the skin. Moreover, newly synthesized collagen may alter the irregular pattern of the connective tissue responsible for the formation of cellulite.

ELIGIBILITY:
Inclusion Criteria:

* Areas for which cellulite appearance reduction is being sought are the bilateral thighs and buttocks
* Clinical cellulite gradation of Stage II or III on the Nurnberger-Muller scale for each treatment area
* PI or P2 on the American Society of Anesthesiologists (ASA) Physical Status Classification System
* Willing and able to abstain from partaking in any treatment other than the study procedure to promote cellulite appearance reduction/body contouring/weight loss during the study
* Willing and able to maintain regular diet and exercise regimen without effecting significant change in either direction during the study
* Willing and able to maintain regular medication schedule, as is medically feasible, during the study

Exclusion Criteria:

* Clinical cellulite gradation of Stage 0 or I on the Nurnberger Muller Scale (NMS) for either one or both thighs/buttocks
* P3 or P4 or P5 or P6 on the ASA Physical Status Classification System
* Weight fluctuation greater than 10 pounds in the prior month
* Previous attempt(s) to reduce cellulite in the study treatment areas over the past 6 months
* Prior surgical intervention to the treatment areas, for any reason
* Medical, physical or other contraindications for cellulite reduction/body contouring/weight loss
* Current use of medication(s) known to affect weight levels and/or cause bloating or swelling and for which abstinence during the study is not safe or medically prudent
* Any medical condition known to affect weight levels, cause bloating or swelling
* Diagnosis of, and/or taking medication for, irritable bowel syndrome
* Active infection, wound or other external trauma to the study treatment areas
* Dermatitis or significant scarring in the study treatment areas
* Medical, physical, or other contraindications for, or known sensitivity to, light therapy
* Diabetes dependent on insulin or oral hypoglycemic medications
* Known cardiovascular disease
* Cardiac surgeries
* History of deep venous thrombosis, arterial disease of the legs
* Pregnant, breast feeding, or planning pregnancy prior to study end
* Serious mental health illness or psychiatric hospitalization in past 2 years
* Developmental disability or cognitive impairment that would impact study participation
* Involved in litigation/receiving disability benefits related to the parameters of the study
* Participation in research in the past 30 days

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Roche, D.O., Principal Investigator; Robert F Jackson, M.D., Principal Investigator
Locations (2):
- United States (2):
  - Surgeon's Inc., Marion, Indiana
  - Bloomfield Laser and Cosmetic Surgery Center, Bloomfield Hills, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Erchonia Scanner Device (GLS): The Erchonia® GLS device is made up of six independent diodes, each emitting 17 mW, 532 nanometer of green laser light.
  Erchonia Scanner device (GLS): The Erchonia® GLS device is made up of six independent diodes, each emitting 17 mW, 532 nanometer of green laser light.
- Total: Total of all reporting groups
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.87 (10.08) | 39.94 (10.72) | 39.91 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 31 | 31 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68
Stage on the Nurnberger-Muller Scale (NMS) [Number; unit: participants] — The Nurnberger-Muller Scale (NMS) is a four-stage scale to classify stage or degree of cellulite. Stage II is defined as dimpling appearing spontaneously when standing but not when lying down. Orange peel appearance of the skin is evident to the naked eye without need for manipulation. Stage III is defined as dimpling spontaneously present with standing and lying down, evident to the naked eye without manipulation. Orange peel skin surface appearance with raised areas and nodules. NMS is assessed for both legs of each participant, and the worse of the stages is reported.
  participants
    Stage II | 19 | 18 | 37
    Stage III | 15 | 16 | 31
Circumference measurement [Mean (Standard Deviation); unit: inches] — Circumference of the upper right and left thighs was recorded in inches (ins) using a flexible tape measure at standardized measurement points. Results are reported as combined bilateral (right+left thigh) circumference measurements.
  inches | 47.09 (3.65) | 46.05 (4.66) | 46.55 (3.92)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Measured as kilograms per meter squared (kg/m2)
  kg/m2 | 25.42 (2.84) | 24.98 (2.77) | 25.22 (2.80)
Percent Total Body Surface Area (TBSA) [Mean (Standard Deviation); unit: percentage of TBSA] — The % Total Body Surface Area (% TBSA) covered by cellulite was marked and quantified according to the Lund and Browder Chart and methodology. The Lund and Browder chart is widely considered the most accurate method of determining Body Surface Area (BSA). It consists of an anterior and posterior diagram of a patient that is divided into sections. The % TBSA is the sum of the marked areas. The % TBSA of the buttocks and bilateral thighs area, front and back combined, affected by cellulite was calculated according to the Lund and Browder Chart.
  percentage of TBSA | 15.52 (6.06) | 14.38 (7.01) | 14.87 (6.54)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Met the Individual Success Criteria
Description: The individual subject success was defined as a decrease of one or more stages on the Nurnberger-Muller Scale (NMS) from baseline to 2 weeks post-assessment for both of the right and left thighs. The NMS is a four-stage scale used as an industry standard to classify stage or degree of cellulite and to determine change in stage or degree of cellulite following treatment intervention. The NMS ranges from Stage 0 (no cellulite) to Stage III (worse cellulite). A decrease in NMS Stage indicates reduced appearance of cellulite and is positive for study success. An increase in NMS Stage indicates worsened appearance of cellulite and is negative for study success. Overall study success was defined as 35% more subjects in the test group than in the control group attaining individual subject success. Results are reported below as the number of subjects in each group that met the individual subject success criteria.
Time Frame: Baseline and 2 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device
Number analyzed (Participants) | 34 | 34
participants | 19 | 3
Statistical Analysis 1: Comparison: Erchonia Scanner Device (GLS) vs Placebo Device; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Bilateral Upper Thigh Circumference Measurement
Description: Circumference of the upper right and left thighs was recorded in inches (ins) using a flexible tape measure and the two measurements were summed, at baseline and 2 weeks. A decrease in bilateral upper thigh circumference measurements is positive in support of study success and an increase in bilateral circumference measurements is negative in support of study success.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device
Number analyzed (Participants) | 34 | 34
inches | -0.85 (1.01) | -0.39 (0.71)
Statistical Analysis 1: Comparison: Erchonia Scanner Device (GLS) vs Placebo Device; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Change in Body Weight
Description: Body weight is measured in pounds (lbs) using a digital scale.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device
Number analyzed (Participants) | 34 | 34
pounds | -1.41 (1.62) | -0.31 (1.59)
Statistical Analysis 1: Comparison: Erchonia Scanner Device (GLS) vs Placebo Device; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

4. Secondary Outcome: Change in Percent (%) Body Surface Area (BSA) Covered by Cellulite.
Description: The % Total Body Surface Area (% TBSA) covered by cellulite was marked and quantified according to the Lund and Browder Chart and methodology. The Lund and Browder chart is widely considered the most accurate method of determining Body Surface Area (BSA). It consists of an anterior and posterior diagram of a patient that is divided into sections. The % TBSA is the sum of the marked areas. The % TBSA of the buttocks and bilateral thighs area, front and back combined, affected by cellulite was calculated according to the Lund and Browder Chart.
Time Frame: Baseline and 2 weeks
Population: The number of subjects analyzed for % TBSA covered by cellulite is less than the total number enrolled as this measure was not recorded for all subjects.
Measure: Mean (Standard Deviation); unit: percentage of TBSA
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device
Number analyzed (Participants) | 23 | 29
percentage of TBSA | -3.89 (1.45) | -0.66 (0.23)
Statistical Analysis 1: Comparison: Erchonia Scanner Device (GLS) vs Placebo Device; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

5. Secondary Outcome: Patient Satisfaction With Study Outcome
Description: At completion of the treatment administration phase, the subject was asked to indicate how satisfied he or she was with any overall perceived change in the appearance of cellulite in his or her thighs and buttocks using the following five-point scale:
  Very Satisfied Somewhat Satisfied Neither Satisfied nor Dissatisfied Not Very Satisfied Not at All Satisfied
  Results are reported as the number of subjects who reported being 'Very Satisfied' or 'Somewhat Satisfied' with the study outcome.
Time Frame: 2 Weeks
Measure: Number; unit: participants
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device
Number analyzed (Participants) | 29 | 31
participants | 18 | 8

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Erchonia Scanner Device (GLS) | Placebo Device
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No